CLINICAL TRIAL: NCT02301078
Title: Comparing Short-term Function and Pain After Treatment With Collagenase Clostridium Histolyticum or Percutaneous Needle Aponeurotomy for Dupuytren's Disease
Brief Title: Short-term Function and Pain After Treatment for Dupuytren's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Other Study IDs: Pain and Function - PNA vs CCH
Record Dates: First submitted 2014-07-11; First posted 2014-11-25 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Dupuytren Disease
Keywords: Dupuytren disease; needle aponeurotomy; collagenase
MeSH Terms: conditions — Dupuytren Contracture | interventions — Fasciotomy; Microbial Collagenase

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Percutaneous Needle Aponeurotomy: Patients who choose to undergo percutaneous needle aponeurotomy (PNA) for primary treatment of Dupuytren's disease
  Interventions: Procedure: Percutaneous Needle Aponeurotomy
- Xiaflex: Patients who choose to receive Collagenase clostridium histolyticum injection (drug name Xiaflex) for primary treatment of Dupuytren's disease.
  Interventions: Drug: Collagenase clostridium histolyticum

INTERVENTIONS:
Procedure: Percutaneous Needle Aponeurotomy — single procedure (day 0)
  Other Names: needle aponeurotomy; fasciotomy
  Groups: Percutaneous Needle Aponeurotomy
Drug: Collagenase clostridium histolyticum — Xiaflex injection into palpable cords (day 0), physical manipulation (day 7)
  Other Names: Xiaflex
  Groups: Xiaflex

SUMMARY:
This study will evaluate short-term pain and function associated with percutaneous needle aponeurotomy (PNA) and injections of the enzyme collagenase clostridium histolyticum in patients with Dupuytren's disease. Scores on outcome measures will be compared between groups to determine whether treatments differ in terms of hand function and pain during the early post-treatment period.

DETAILED DESCRIPTION:
Percutaneous needle aponeurotomy (PNA) and injections of the enzyme collagenase clostridium histolyticum are two non-invasive treatment options for patients with Dupuytren's disease. While PNA has been offered for decades, injectable collagenase is relatively new. The effectiveness of each treatment has been compared in the literature; however, recovery, in terms of pain and short-term function has not been formally evaluated. The objective of this study is to objectively compare short-term function and pain outcomes associated with each of these two procedures in patients presenting with untreated Dupuytren's disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* Dupuytren's disease diagnosis
* Consented to either percutaneous needle aponeurotomy or Xiaflex injection (patient choice)
* Able to read/write/speak English
* Must have an email address

Exclusion Criteria:

* Previous treatment for Dupuytren's disease
* Type 2 Diabetes Mellitus
* Pre-existing hand condition, previous hand surgery or trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at Sunnybrook Health Sciences Centre choosing either percutaneous needle aponeurotomy or Xiaflex injection for treatment of Dupuytren's disease.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-10 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Brief Michigan Hand Questionnaire (brief MHQ) | Baseline
  A validated patient-reported 12-item questionnaire pertaining to several aspects of hand function that is answered on 1 through 5 Likert scales. Higher scores indicate better hand function.
Unite Rhumatologique des Affections de la Main (URAM) scale | Baseline
  The URAM is a validated patient-reported 9-item functional assessment scale used clinically and for research purposes specific to patients with Dupuytren's disease. The resulting score quantifies Dupuytren's disease-related disability, with higher scores indicating higher level of disability.
Daily Pain and Function Scales | Baseline
  An emailed form asking participants to rate pain and function during the past 24 hours using two 1-5 Likert scales. Two additional questions to assess night splint compliance and pain medication (yes/no)
Brief Michigan Hand Questionnaire (brief MHQ) | Day 7
Brief Michigan Hand Questionnaire (brief MHQ) | Day 14
Brief Michigan Hand Questionnaire (brief MHQ) | Day 21
Brief Michigan Hand Questionnaire (brief MHQ) | Day 28
Unite Rhumatologique des Affections de la Main (URAM) scale | Day 7
Unite Rhumatologique des Affections de la Main (URAM) scale | Day 14
Unite Rhumatologique des Affections de la Main (URAM) scale | Day 21
Unite Rhumatologique des Affections de la Main (URAM) scale | Day 28
Daily Pain and Function Scales | Day 1
Daily Pain and Function Scales | Day 2
Daily Pain and Function Scales | Day 3
Daily Pain and Function Scales | Day 4
Daily Pain and Function Scales | Day 5
Daily Pain and Function Scales | Day 6
Daily Pain and Function Scales | Day 7
Daily Pain and Function Scales | Day 14
Daily Pain and Function Scales | Day 21
Daily Pain and Function Scales | Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Division of Plastic and Reconstructive Surgery, Toronto, Ontario, Canada